CLINICAL TRIAL: NCT02465463
Title: A Pilot Study Examining the Safety and Efficacy of Early Fecal Transplant in Patients Infected With Clostridium Difficile at High Risk of Relapse
Brief Title: Early FMT for C.Difficile
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Tanvi Dhere, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00077804
Record Dates: First submitted 2014-11-27; First posted 2015-06-08 (Estimated); Results first posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Clostridium Difficile
Keywords: fecal microbiota transplant; probiotic
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT arm (Experimental): Patients in the experimental arm with undergo a fecal microbiota transplant (FMT) after finishing a course of antibiotics.
  Interventions: Procedure: Fecal microbiota transplant (FMT); Device: flexible sigmoidoscopy
- Control (No Intervention): Patients in the non-interventional group will not receive a FMT but will be followed over the course of 6 months to assess for recurrence of C.difficile.

INTERVENTIONS:
Procedure: Fecal microbiota transplant (FMT) — 250 mL of donor stool will be infused into the colon by flexible sigmoidoscopy
  Arms: FMT arm
Device: flexible sigmoidoscopy
  Arms: FMT arm

SUMMARY:
Clostridium difficile infection (CDI) has increased worldwide in both frequency and severity. It is the leading cause of hospital acquired infection in developed countries and has been associated with at least 14,000 deaths per year in the United States. With 3 million cases/ year, the annual cost for treating the infection is exceeding 3 billion dollars. It can also have a profound negative impact on quality of life.

The investigators believe that patients who are at high risk of relapse after a first CDI episode would benefit from early fecal microbial transplant (FMT). The proposed study will produce preliminary data regarding safety and efficacy and potential for cost effectiveness for the use of early fecal transplant in those patients with their first episode of non-refractory CDI who are predicted to have a high rate of recurrence based on previously published risk factors. The investigators will be better prepared to test the efficacy of this approach in a future multicenter clinical trial in a randomized controlled fashion.

The purpose of this study is to compare the effectiveness and safety of early fecal transplant using donor stool from a healthy person in a group of patients who are diagnosed with their first episode of Clostridium difficile infection and are predicted to have a high chance of the infection returning against a similar group of patients who receive current standard of care for treatment of C.difficile.

The investigators hypothesize:

* that clinical remission rates at 12 weeks as noted by absence of clinical symptoms and/or negative C.difficile stool polymerase chain reaction (PCR) will be greater in the experimental arm compared to the control arm
* that patients in the experimental group will have a low microbial diversity prior to FMT but will exhibit a high microbial diversity after the FMT that resembles the respective donor
* that the microbial diversity will be diminished in both groups at the time of enrollment, but the experimental group will exhibit a higher microbial diversity compared to the control population at 12 weeks
* that patients in both groups will exhibit poor quality of life at the time of enrollment, however, the experimental group will demonstrate higher quality of life compared to the control group at follow up after completion of treatment
* that costs incurred by the experimental group will be less than the control group

DETAILED DESCRIPTION:
Treatment of CDI remains challenging, especially in those with recurrent disease. Failures rates of 20-30% with initial treatment have been reported, and up to 65% fail after a third course of antibiotics. In addition, costs of treatment, which can be upward of $3000 for a 10 day course of a single antibiotic, may leave many patients and their families financially overburdened. Use of FMT has shown to be effective with cure rates above 80%, safe even in immunocompromised patients, and cost effective in those with recurrent (3 or more) episodes of C.difficile. Emory University and Emory Clinic have performed over 100 FMT's since July 2012 for treatment of recurrent or refractory CDI and has had similar cure rates.

Current treatment approaches for CDI limit the use of fecal transplant to those who have had more than 2 recurrences with at least one failure of a 6-8 week taper with vancomycin or at least 2 episodes of severe CDI resulting in hospitalization or refractory CDI defined as moderate CDI not responding to standard therapy for at least one week (5). However, the investigators feel that by attempting to perform FMT early after a first episode in those at high risk of recurrence, decreased recurrence rates, improved quality of life, and lower health care costs will be seen.

Patients who participate will be randomized to one of two groups - one group who receives a fecal transplant and another group who will not receive a fecal transplant. A fecal transplant using a sigmoidoscopy will occur after the subjects in the fecal transplant arm complete the course of antibiotics for treatment of the C.difficile infection. Healthy stool from a donor will be infused into the colon to help replenish good bacteria that patients with C.difficile infection often do not have. The group that does not undergo FMT will take antibiotics and probiotic therapy for management of CDI as part of standard of care.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for the study:

* First or second episode of CDI responding to therapy
* Must have 2 or more of the following criteria:

  1. Age >65
  2. Severe underlying disease (measured by Horn index score of 3 or 4)
  3. Additional non-C.difficile antibiotic exposure during CDI episode
  4. Use of antacids
  5. Previous episode of CDI
* Willingness to accept a fecal product made using unrelated donor stool and to comply with study protocol requirements
* Able to give informed consent
* Chronic infection with HIV, HBV, HCV is permitted unless the viral infection compromises the ability of the patient to safely participate in the study. Patients with a CD4 count <200 and/ or AIDS defining illness or decompensated cirrhosis will not be eligible for the study.
* Life expectancy >4 months

Exclusion Criteria:

* Any of the following: acute leukemia, history of allogenic or recent (within 6 months) autologous bone marrow transplant, or use of cytotoxic chemotherapy within 2 months
* ANC <1000/mm^3
* History of inflammatory bowel disease
* History of total colectomy
* Pregnant or nursing mothers
* History of significant food allergy to foods not excluded from the donor diet
* Patient has any other condition that, in the opinion of the Investigator, would jeopardize the safety or rights of the subject participating in the study, would make it unlikely for the subject to complete the study, or would confound the results of the study
* Patients who are aged 80 years or greater
* Patients who are incarcerated
* Patient with cognitive impairment or severe neuropsychiatric co morbidities who are incapable of giving consent
* Inherited/primary immune disorders
* Patients who are unwilling or unable to undergo sigmoidoscopy
* Unable to comply with protocol requirements
* Patients with untreated, in-situ colorectal cancer

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanvi Dhere, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited June 2015 through November 2016.
Groups:
- FMT Arm: Patients in the experimental arm underwent a fecal microbiota transplant (FMT) after finishing a course of antibiotics.
  Fecal microbiota transplant (FMT): 250 mL of donor stool was infused into the colon by flexible sigmoidoscopy
  flexible sigmoidoscopy
- Control: Patients in the non-interventional group did not receive a FMT but were followed over the course of 6 months to assess for recurrence of C.difficile.
Period: Overall Study
Arm/Group | FMT Arm | Control
Started | 8 | 5
Completed | 4 | 4
Not Completed | 4 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants that have completed the study.
Groups:
- FMT Arm: Patients in the experimental arm with undergo a fecal microbiota transplant (FMT) after finishing a course of antibiotics.
  Fecal microbiota transplant (FMT): 250 mL of donor stool will be infused into the colon by flexible sigmoidoscopy
  flexible sigmoidoscopy
- Total: Total of all reporting groups
Arm/Group | FMT Arm | Control | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.25 (9.34) | 61.75 (7.20) | 59.13 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission Rates
Description: Clinical remission rate is defined as the number of participants with an absence of clinical symptoms and/or negative C.difficile stool PCR.
Time Frame: Post-Intervention (Week 12)
Population: Participants that completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- FMT Arm: Patients in the experimental arm will undergo a fecal microbiota transplant (FMT) after finishing a course of antibiotics.
  Fecal microbiota transplant (FMT): 250 mL of donor stool will be infused into the colon by flexible sigmoidoscopy
  flexible sigmoidoscopy
Arm/Group | FMT Arm | Control
Number analyzed (Participants) | 4 | 4
Participants | 3 | 2

2. Primary Outcome: Number of Participants That Experience Serious Adverse Events
Description: A serious adverse event is any adverse experience that results in any of the following outcomes:
  * Death;
  * Life-threatening experience (adverse event is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death);
  * Requires inpatient hospitalization or prolongation of existing hospitalization;
  * Results in persistent or significant disability or incapacity;
  * Is a congenital anomaly or birth defect;
  * Is considered to be an important medical event (that may not be immediately life threatening or result in death or hospitalization but may jeopardize the patient or may require intervention to prevent one of the outcomes listed in the definition above).
Time Frame: Post-Intervention (Month 6)
Population: Participants that completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Arm | Control
Number analyzed (Participants) | 4 | 4
Participants | 0 | 0

3. Primary Outcome: Change in the Shannon Diversity Index
Description: The Shannon Diversity Index is a quantitative measure that reflects how many different types (such as species) there are in a dataset (a community). 16s ribosomal gene sequencing and metabolomic profile of the gut microbiota were analyzed for both groups using the Shannon Diversity index (H). The greater the index, the more diverse a species.
Time Frame: Baseline, Post-Intervention (Week 12)
Population: Participants that completed the study.
Measure: Number; unit: H
Arm/Group | FMT Arm | Control
Number analyzed (Participants) | 4 | 4
H
  Baseline | 2.46 | 2.22
  Post-Intervention (Week 12) | 2.55 | 2.34

4. Secondary Outcome: Mean Short Form - 36 (SF-36) Score
Description: SF-36: consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Post-Intervention (Week 12)
Population: Participants that have completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FMT Arm | Control
Number analyzed (Participants) | 4 | 3
units on a scale | 89.93 (9.8) | 52.71 (25.78)

5. Secondary Outcome: Mean Hospital Anxiety And Depression Scale (HADS) Score
Description: The HADS is a fourteen item scale and each item on the questionnaire is scored from 0-3, from 0 = best and 3 = worst. A score can range between 0 and 21 for either anxiety or depression. Higher scores represent greater depressive/anxious symptoms.
Time Frame: Post-Intervention (Week 12)
Population: No difference in anxiety and depression scores were seen between the two populations at baseline and at 12 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FMT Arm | Control
Number analyzed (Participants) | 4 | 3
units on a scale | 3 (3.56) | 5.67 (4.51)

6. Secondary Outcome: Mean Cost of Treatment
Description: Total cost was calculated as a summation of costs of medications, procedures, and fecal transplant used to treat C.difficile for each individual patient. A mean was calculated for both groups.
Time Frame: Post-Intervention (Month 6)
Population: Participants that have completed the study.
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | FMT Arm | Control
Number analyzed (Participants) | 4 | 4
dollars | 543.6 (0) | 1481.7 (1780.79)

ADVERSE EVENTS:
Arm/Group | FMT Arm | Control
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No